CLINICAL TRIAL: NCT01992250
Title: Freezing Alone Instead of Resection Of Small Breast Tumors: A Study of Cryoablation in the Management of Early Stage Breast Cancer
Brief Title: Cryoablation of Small Breast Tumors in Early Stage Breast Cancer
Acronym: FROST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sanarus Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-00-0011
Record Dates: First submitted 2013-11-06; First posted 2013-11-25 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
Keywords: Cryoablation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Risk - Age 70+ (Other): Age 70+. Patients treated with the Visica 2 Treatment System, followed by adjuvant therapies
  Interventions: Device: Visica 2 Treatment System
- Moderate Risk - Age 50-69 (Other): Age between 50-69. Patients treated with the Visica 2 Treatment System, followed by adjuvant therapies
  Interventions: Device: Visica 2 Treatment System

INTERVENTIONS:
Device: Visica 2 Treatment System — Cryoablation
  Other Names: Visica Breast Therapy

SUMMARY:
This study examines the use of cryoablation as an alternative to surgery in the treatment of early stage invasive breast cancer. The hypothesis is that cryoablation will complete ablation and destroy the tumor in a selected population of women who may otherwise be adequately treated with surgery.

DETAILED DESCRIPTION:
PURPOSE:

To determine the rate of successful tumor ablation in patients treated with cryoablation and endocrine therapy in a subset of patients with early stage breast cancer.

OUTLINE:

1. Core Biopsy (Pre-Registration)
2. Magnetic Resonance Imaging (Pre-Registration)
3. Tumor Cryoablation
4. Core Biopsy (Post-Cryoablation)
5. Magnetic Resonance Imaging (Post-Cryoablation)
6. Postoperative Follow-up
7. Evaluation of outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50
2. Unifocal primary invasive breast carcinoma diagnosed by core needle biopsy
3. Maximum tumor size ≤1.5 cm in its greatest diameter
4. Ultrasound visible lesion(s)
5. Clinically node negative, hormone receptor positive (+). HER2 negative (-), with <25% intraductal component in the aggregate.
6. Unilateral or bilateral disease meeting study criteria
7. Physical and emotional ability to undergo baseline and follow-up breast MRIs and serial breast cosmesis analysis
8. Patient agrees to receive a 5 year minimum course of endocrine therapy following cryoablation for control of systemic disease

Exclusion Criteria:

1. Prior treatment (e.g., open surgical biopsy, lumpectomy) of index cancer
2. Ductal carcinoma in-situ with microinvasions (T1mic)
3. Multifocal or multicentric invasive breast carcinoma
4. Prior or planned neoadjuvant systemic therapy for breast cancer
5. Tumor with ≥25% IDC components

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-11; Primary Completion 2021-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Tumor ablation occurence | Within 6 months
  Successful tumor ablation will be defined as absence of residual viable invasive or in situ carcinoma. Will be determined at 6-month post-cryoablation biopsy. Residual disease will require surgery.

SECONDARY OUTCOMES:
Local tumor recurrence | Within 5 years
Satisfactory breast cosmesis results | 5 Years
Adverse event assessment | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dennis R. Holmes, MD, FACS, Principal Investigator — 90210 Surgery Medical Center
Locations (12):
- United States (12):
  - Arizona Breastnet, Scottsdale, Arizona
  - 90210 Surgery Medical Center, Beverly Hills, California
  - City of Hope, Duarte, California
  - Epic Care, Emeryville, California
  - Diagnostic Center for Women, LLC, Miami, Florida
  - Naples Community Hospital, Naples, Florida
  - Ascension Crittenton Hospital, Rochester, Michigan
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Knoxville Comprehensive Breast Center, Knoxville, Tennessee
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Ogden Regional Hospital, Ogden, Utah

IPD SHARING:
Plan to Share IPD: Undecided